CLINICAL TRIAL: NCT02534311
Title: Prospective Evaluation of Rheumatoid Arthritis Activity Using DAS28 in Patients Treated With Subcutaneously Administered Tocilizumab on Local Level
Brief Title: A Phase IV Study to Evaluate the Effect of Subcutaneous (SC) Tocilizumab Administered to Participants With Rheumatoid Arthritis (RA) Assessed Using Disease Activity Score (DAS28)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29712
Record Dates: First submitted 2015-08-25; First posted 2015-08-27 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Tocilizumab: Participants will receive tocilizumab (162 milligrams [mg]) SC injection for 48 weeks.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab will be administered at 162 mg SC injection for 48 weeks.
  Other Names: RoActemra

SUMMARY:
The purpose of this clinical trial is to prospectively evaluate RA activity using the assessment of change in DAS28 under local conditions in Slovakia in participants who are treated with subcutaneously administered tocilizumab pursuant to the recommendations of the Ministry of Health of the Slovak Republic in order to better assess the disease activity and impairment of the joint function.

ELIGIBILITY:
Inclusion Criteria:

* Participants with age greater than or equal to (>=) 18 years
* Participants with moderate to severe active RA (DAS28 >=3.2) who did not respond sufficiently to or did not tolerate previous treatment with one or several disease-modifying antirheumatic drugs (DMARDs), irrespective of whether they were of biological or synthetic nature
* Participants eligible for the treatment with subcutaneously administered tocilizumab, as decided by the doctor in accordance with summary of product characteristics (SPC) and standard therapeutic procedures, who were not previously treated with tocilizumab and did not receive any other biological treatment for RA in the past either
* Assignment of participants for observation using the treatment described above is clearly separated from the physician's decision to prescribe the treatment to the patient.
* Pulmonologist's consent for chest X-ray and quantiferon test with commencement of biological treatment

Exclusion Criteria:

* Hepatitis B surface antigen (HBsAg,) hepatitis C virus (HCV) or human immunodeficiency virus (HIV) positivity
* History of severe allergic or anaphylactic responses to human or humanized murine monoclonal antibodies
* History of intestinal ulcerations or diverticulitis
* Active hepatopathy with more than threefold increase of alanine transaminase (ALT) or aspartate transaminase (AST)
* Thrombocytes <100,000 per cubic milliliters (/mm^3), less than (<) 3,000 mm^3, absolute neutrophil count < 2,000 mm^3
* Women of childbearing age (without medically confirmed sterility, e.g. following hysterectomy, ovariectomy, menopause lasting 2 years) who do not accept the use of a suitable form of contraception (e.g. barrier methods of contraception in the participant and partner, contraceptive pills or patches, hormonal implants, spermicidal agents in combination with barrier method of contraception, intrauterine device)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Moderate to severe RA participants who are treated with tocilizumab
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-10-13 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2015-12-01 (Actual)

PRIMARY OUTCOMES:
Average change from baseline in DAS28 | up to Week 24
Average change from baseline in DAS28 | up to Week 48

SECONDARY OUTCOMES:
Percent of participants achieving clinical remission defined as a DAS28 <2.6 | Baseline, Week 12, 24, 36, and 48
Percentage of participants achieving a DAS28 >=3.2 | Baseline, Week 12, 24, 36, and 48
Evaluation of participant's pain using visual analogue scale (VAS) | Baseline, Week 12, 24, 36, and 48
Evaluation of the disease activity by participant using VAS | Baseline, Week 12, 24, 36, and 48
Evaluation of the disease activity by Doctor using VAS | Baseline, Week 12, 24, 36, and 48
DAS28-joint count (erythrocyte sedimentation rate) [DAS28(ESR)] score | Baseline, Week 12, 24, 36, and 48
DAS28-joint count (C-reactive protein) [DAS28(CRP)] score | Baseline, Week 12, 24, 36, and 48
Absolute and percent change in the Health Assessment Questionnaire (HAQ) | Baseline, Week 12, 24, 36, and 48

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- Slovakia (4):
  - Banská Bystrica
  - Bratislava
  - Nitra
  - Piešťany